CLINICAL TRIAL: NCT04172935
Title: Productivity Study of Presbyopia Improvement in Textile Workers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSU-OPH-005
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Presbyopia
Keywords: Presbyopia; textile worker
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Presbyopic Glasses/ Intervention Group (Experimental): Immediate provision of a free pair of spherical presbyopic glasses to correct the worker's vision for optimal working distance as measured before intervention.
  Interventions: Device: Presbyopic Glasses/ Intervention Group
- Control Group (No Intervention): Will be deferred to receive spectacles as above, after the 4 weeks evaluation period.

INTERVENTIONS:
Device: Presbyopic Glasses/ Intervention Group — Immediate provision of a free pair of spherical presbyopic glasses to correct the worker's vision for optimal picking distance, astigmatism is corrected.
  Arms: Presbyopic Glasses/ Intervention Group

SUMMARY:
To establish, using a randomized, controlled design, the impact of near vision correction on the productivity of presbyopic textile workers in China, as measured by the change of monthly income.

DETAILED DESCRIPTION:
Sustainable development is considered to be a major development strategy to meet rapid economic and social development in China. China is one of the biggest manufacturing hubs in the world. With the rapid development of economy, the health of manufacturing workers is closely related to productivity. In some low-income developing countries, studies have focused on improving the health of manufacturing workers to improve productivity .Most of the studies focused on improving the nutritional intake of workers has a significant effect on improving work efficiency and productivity .

As the global aging is becoming an critical issue for both health and economics, the health of the working population over the age of 45 is of greater concern in low - and middle-income developing countries. China has a workforce of 980 million people (aged 15 to 60). Urban workers and blue-collar workers account for nearly 310 million. With the aging population increased, presbyopia is becoming more and more serious, and it also affects the labor group that needs to work in close proximity. Studies have proved that refractive correction for tea pickers with old vision can effectively improve the yield of tea pickers and increase personal income.Because Guangdong area textile industry is developed, textile worker population is large. Most front-line textile workers need to work in close proximity for a long time, and the problem of aging productivity is increasingly obvious. At present, no relevant studies have explored whether presbyopia affects the work efficiency of textile workers who work in close proximity.

In this study, a randomized controlled clinical study will be conducted on front-line textile workers with presbyopia to explore whether refractive correction can improve labor income and relieve symptoms of visual fatigue for textile workers aged 40 years or above who work in the front-line.

ELIGIBILITY:
Inclusion Criteria:

* Employee of E-square for 6 months;
* Aged >= 40 years;
* Quantifiable near visual task workers;
* Habitual near visual acuity of >= 0.8M (<=6/12) at 40cm in both eyes, correctable to <=0.5M (>=6/7.5);
* Near correction spherical equivalent refractive error >= +0.50D or astigmatism <-1.00D;
* Asthenopia symptoms reported ( Asthenopia questionnaire score >= 16) Ability to give informed consent

Exclusion Criteria:

* Ocular surgery done in the past 3 months;
* Eye disease detected on baseline eye exam
* Current ownership of near correction capable of improving near visual acuity to <= 0.8M (>= 6/12) in either eye
* Unlikely to complete follow-up due to unsatisfactory work performance, plans to move out of the area, etc.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2019-12-13 (Estimated); Primary Completion 2019-12-21 (Estimated); Study Completion 2049-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of income change of textile workers | 4 weeks
  The rate of income change over baseline.

SECONDARY OUTCOMES:
The quality of vision function | 4 weeks
  Secondary outcome will be the quality of vision function in both groups.National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25 ) questionnaire will be used to measure the quality of vision function.For the NEI-VFQ-25, a composite score (25 items) and near activities sub score (two items) were created on 0-100 scales.
Percentage of glasses wear in intervention group, as well as the purchase and use of glasses in control group. | 4 weeks
  Independent compliance observation of wear of the study spectacles in the intervention group, self-reported purchase and use of glasses in the control group will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yangfa Zeng, Master, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Gaoming, Foshan, Guangdong, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No